CLINICAL TRIAL: NCT05119413
Title: Comparison of a New Masterful Preparation to Kligman's Trio in the Treatment of Melasma: a Double Blind Prospective Randomzed Study
Brief Title: Comparison of a New Masterful Preparation to Kligman's Trio in the Treatment of Melasma
Acronym: Kligman
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-PP-30
Record Dates: First submitted 2021-10-04; First posted 2021-11-15 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New traitement (Experimental): Thiamidol, retinoid, topical steroid preparation
  Interventions: Drug: New trio de Kligman
- Kligman's trio (Other): Application once a day for 12 weeks
  Interventions: Drug: Trio Kligman

INTERVENTIONS:
Drug: New trio de Kligman — Once daily application in addition to the same sunscreen
  Arms: New traitement
Drug: Trio Kligman — Once daily application in addition to the same sunscreen
  Arms: Kligman's trio

SUMMARY:
Kligman's trio remains the gold standard treatment for melasma. It contain hydroquinone which is an effective anti-melanogenic compound but that has poor tolerance and numerous side-effects. Thiamidol has been proven to be at least as effective as hydroquinone and has a very good safety profile. The objective of this study is to compare the Kligman's trio to the same preparation in which hydroquinone is replaced by thiamidol.

ELIGIBILITY:
Inclusion Criteria:

* SIGNED WRITTEN CONSENT 1) Melasma clinically diagnosed

Exclusion Criteria:

1. Pregnant woman
2. Other pigmentary disorder affecting the face
3. Use of systemic or topical steroids or retinoids, use of topical depigmenting agents or depigmenting procedure in the month before the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The melasma's type | at 12 weeks
  Clinical score MASI

SECONDARY OUTCOMES:
the Quality of life of patient | at 12 weeks
  descriptive name of scale : meslascol

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No